CLINICAL TRIAL: NCT04004325
Title: A Phase 1/2, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability and Efficacy of FT-4101 in Overweight/Obese Subjects With NASH
Brief Title: A Study of FT 4101 in Overweight/Obese Participants With Non-alcoholic Steatohepatitis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Forma Therapeutics, Inc. (Industry)
Collaborators: ProSciento, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4101-MET-201
Record Dates: First submitted 2019-06-10; First posted 2019-07-02 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Nonalcoholic Steatohepatitis (NASH); Overweight or Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental)
  Interventions: Drug: FT-4101; Drug: FT-4101 placebo; Other: Deuterated Water
- Cohort B (Experimental)
  Interventions: Drug: FT-4101; Drug: FT-4101 placebo; Other: Deuterated Water

INTERVENTIONS:
Drug: FT-4101 — FT-4101 will be supplied as active capsules and will be administered per the protocol defined frequency and dose level.
Drug: FT-4101 placebo — FT-4101 placebo will be supplied as placebo capsule matching in size and color to all the active capsules and will be administered per the protocol defined frequency and dose level.
Other: Deuterated Water — Deuterated water will be provided as individual ready-to-use, single dose bottles each containing 50 mL of deuterated water (70%).

SUMMARY:
This Phase 1/2 study will evaluate safety, efficacy, PK, and PD of FT-4101 as a single agent in overweight/obese subjects with NASH.

The study may be conducted in up to 2 dosing cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Meets all of the following criteria:

  1. CAP ≥ 300 dB/m by FibroScan® OR Liver biopsy within 24 months, consistent with NASH with stage 2-3 fibrosis
  2. Screening MRI-PDFF with ≥ 10% steatosis.
* Body mass index (BMI) > 25.0 to < 45.0 kg/m2
* Stable body weight
* Subjects with T2DM may also be included, if:

  1. Subject with T2DM is on stable doses of metformin monotherapy (subjects on combination therapy of metformin and sulfonylurea (SU) need to undergo washout period prior to dosing) with no changes in medication within the previous 6 months
  2. HbA1c < 9% (one retest is permitted with the result of the last test being conclusive)
  3. Fasting plasma glucose (FPG) < 240 mg/dL (<13.3 mmol/L)
* Waist circumference ≤ 57 inches
* Female subjects must be non-pregnant and non-lactating

Key Exclusion Criteria:

* Type 1 diabetes and type 2 diabetic subjects on insulin therapy
* Diabetic complications, such as acute proliferative retinopathy
* Recurrent severe hypoglycemia or hypoglycemic unawareness or recent severe ketoacidosis
* History of, or active, chronic liver disease due to alcohol, auto-immune, primary biliary cholangitis, HIV, HBV or active HCV-infection, Wilson's, α-1-antitrypsin deficiency, hemochromatosis, etc., and not due to NASH disease
* History of clinically significant or decompensated chronic liver disease including esophageal varices, ascites, encephalopathy or any hospitalization for treatment of chronic liver disease; or MELD score ≥ 10.
* History of significant cirrhosis of the liver
* Alcohol consumption greater than 14 drinks per week for men or greater than 7 drinks per week for women and/or positive alcohol breath test
* Introduction of an anti-obesity drug in the past 6 months prior to screening
* History of gastrointestinal malabsorptive bariatric surgery, any other gastrointestinal surgery that may induce malabsorption, history of bowel resection > 20 cm, any malabsorption disorder, severe gastroparesis, any GI procedure for weight loss, as well as clinically significant gastrointestinal disorders within less than 5 years
* Ingestion of drugs known to produce hepatic steatosis including corticosteroids, high- dose estrogens, methotrexate, tetracycline or amiodarone in the previous 6 months
* History of, or current cardiac dysrhythmias and/or a history of cardiovascular disease events, including congestive heart failure, unstable coronary artery disease, myocardial infarction
* Significant systemic or major illnesses other than liver disease, including cerebrovascular disease, pulmonary disease, renal failure, organ transplantation, serious psychiatric disease, malignancy that, in the opinion of the investigator, would preclude treatment with FT-4101 and/or adequate follow up
* History of chronic skin conditions such as psoriasis, eczema or any recurring rash/dermatitis requiring oral or topical corticosteroids or other topical applications within 12 months
* Hair loss or unexplained alopecia within 12 months
* History of chronic eye conditions, Sjögren syndrome or any history of dry eyes or allergic conjunctivitis requiring artificial tears or medicated eye drops or previous refractive surgery within 12 months (Subjects with dry eyes due to wearing contact lenses are eligible)
* History of major depression, anxiety, suicidal behavior or attempts, or other unstable psychiatric disorders (within 2 years of screening), requiring medical treatment
* Uncontrolled hypertension
* Any device or other contraindication with the MRI examination
* Ingestion of deuterated water within the previous 6 months
* Positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus type 1 (HIV-1) or type 2 (HIV-2) antibody
* Participation in any other clinical interventional study receiving active treatment within the previous 30 days or 5 half-lives, whichever is longer
* Unable to abstain from smoking during confinement periods
* History of illicit drug abuse
* Clinically under the effect of marijuana at screening
* Unwillingness to abstain from grapefruit (grapefruit containing food and beverages), star fruit (carambola), pomegranate, Seville orange and other food components that may interact with CYP3A4 from check-in throughout the entire course of the study
* Donation or loss of > 500 mL of blood or blood product within 56 days of dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), MD, Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - ProSciento, Inc., Chula Vista, California
  - Catalina Research Institute, Montclair, California

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized at a ratio of 2:1 in FT-4101 treatment group and placebo.
Groups:
- FT-4101 3.0 mg: Participants received 3.0 mg of FT-4101 capsule orally once daily for 2 weeks, followed by 1 week of no treatment. This cycle continued until the end of week 12, for up to 4 dosing cycle (each cycle 21 days).
- Placebo: Participants received FT-4101 matching placebo capsule orally once daily for 2 weeks, followed by 1 week of no treatment. This cycle continued until the end of week 12, for up to 4 dosing cycle (each cycle 21 days).
Period: Overall Study
Arm/Group | FT-4101 3.0 mg | Placebo
Started | 9 | 5
Completed | 9 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | FT-4101 3.0 mg | Placebo | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.8 (10.52) | 47.0 (15.76) | 44.9 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 5 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as an adverse events (AEs) with an onset that occurred after receiving the first dose of the study drug (AE start date greater than or equal to [>=] first dose date) and within 30 days after receiving the last dose of the study drug (AE start date - last dose date less than or equal to [<=] 30). Number of participants with TEAEs are reported.
Time Frame: From start of study drug administration up to 20 weeks
Population: The Safety analysis set included all randomized participants who received investigational product (IP) (FT-4101 or placebo) or deuterated water.
Measure: Count of Participants; unit: Participants
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
Participants | 3 | 3

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Values
Description: Number of participants with clinically significant changes in laboratory values (hematology, serum chemistry, and urinalysis) are reported.
Time Frame: Up to 20 weeks
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Count of Participants; unit: Participants
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination
Description: Number of participants with clinically significant changes in physical examination are reported.
Time Frame: Up to 20 weeks
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Count of Participants; unit: Participants
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
Participants | 0 | 0

4. Primary Outcome: Change From Baseline in Vital Signs: Blood Pressure (BP)
Description: Change from baseline in blood pressure (systolic and diastolic) are reported.
Time Frame: Baseline, Day 92
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
millimeters of mercury (mmHg)
  Systolic BP | -0.2 (16.45) | -5.2 (8.44)
  Diastolic BP | 0.4 (14.93) | -2.4 (6.11)

5. Primary Outcome: Change From Baseline in Vital Signs: Heart Rate (HR)
Description: Change from baseline in heart rate is reported.
Time Frame: Baseline, Day 92
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Mean (Standard Deviation); unit: Beats per minutes (beats/min)
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
Beats per minutes (beats/min) | 4.4 (8.32) | 0.2 (2.59)

6. Primary Outcome: Change From Baseline in Vital Signs: Respiratory Rate
Description: Change from baseline in respiratory rate is reported.
Time Frame: Baseline, Day 92
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Mean (Standard Deviation); unit: Breaths per minute (breaths/min)
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
Breaths per minute (breaths/min) | -1.6 (1.42) | -0.6 (1.34)

7. Primary Outcome: Change From Baseline in Vital Signs: Temperature
Description: Change from baseline in temperature is reported.
Time Frame: Baseline, Day 92
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Mean (Standard Deviation); unit: Degree Celsius (C)
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
Degree Celsius (C) | 0.22 (0.239) | -0.08 (0.409)

8. Primary Outcome: Change From Baseline in 12-lead Electrocardiogram (ECG) Parameters: ECG Mean Heart Rate
Description: Change from baseline in ECG mean heart rate is reported.
Time Frame: Baseline, Day 92
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
beats/min | 0.3 (11.46) | 2.6 (6.23)

9. Primary Outcome: Change From Baseline in 12-lead ECG Parameters: QT Interval
Description: Change from baseline in QT interval is reported.
Time Frame: Baseline, Day 92
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
milliseconds (msec) | 0.2 (14.28) | -4.2 (22.80)

10. Primary Outcome: Change From Baseline in 12-lead ECG Parameters: PR Interval
Description: Change from baseline in PR interval is reported.
Time Frame: Baseline, Day 92
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
msec | -7.0 (13.63) | 2.2 (10.64)

11. Primary Outcome: Change From Baseline in 12-lead ECG Parameters: QRS Interval
Description: Change from baseline in QRS interval is reported.
Time Frame: Baseline, Day 92
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
msec | 1.9 (8.62) | 0.8 (8.38)

12. Primary Outcome: Change From Baseline in 12-lead ECG Parameters: RR Interval
Description: Change from baseline in RR interval is reported.
Time Frame: Baseline, Day 92
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
msec | 1.7 (138.73) | -40.8 (93.04)

13. Primary Outcome: Change From Baseline in 12-lead ECG Parameters: QTc (Corrected) Using the Fridericia Correction (QTcF) Interval
Description: Change from baseline in QTcF interval is reported.
Time Frame: Baseline, Day 92
Population: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 9 | 5
msec | 0.6 (10.92) | 1.0 (14.00)

14. Primary Outcome: Percent Change From Baseline in Liver Fat on Magnetic Resonance Imaging- Proton Density Fat Fraction (MRI-PDFF)
Description: Percent change from baseline in liver fat on MRI-PDFF is reported.
Time Frame: At week 12
Population: The preliminary efficacy analysis set included all participants who received FT-4101 or placebo with at least one quantifiable baseline and one post-baseline MRI-PDFF without major protocol deviations or violations that would have an impact on pharmacodynamics (PD) (Specifically MRI-PDFF).
Measure: Mean (Standard Deviation); unit: Percent change of liver fat
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 8 | 5
Percent change of liver fat | -18.02 (20.066) | 25.98 (15.670)

15. Primary Outcome: Change From Baseline in Liver Fat on Magnetic Resonance Imaging- Proton Density Fat Fraction (MRI-PDFF)
Description: Change from baseline in percentage of liver fat on MRI-PDFF is reported.
Time Frame: At week 12
Population: The preliminary efficacy analysis set included all participants who received FT-4101 or placebo with at least one quantifiable baseline and one post-baseline MRI-PDFF without major protocol deviations or violations that would have an impact on PD (Specifically MRI-PDFF).
Measure: Mean (Standard Deviation); unit: Percentage of liver fat
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 8 | 5
Percentage of liver fat | -3.65 (4.389) | 4.16 (2.236)

16. Secondary Outcome: Change From Baseline in Liver Fat on MRI-PDFF
Description: Change from baseline in percentage of liver fat on MRI-PDFF is reported.
Time Frame: At week 6
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percentage of liver fat
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 8 | 5
Percentage of liver fat | -0.10 (3.395) | 3.58 (4.060)

17. Secondary Outcome: Percent Change From Baseline in Liver Fat on MRI-PDFF
Description: Percent change from baseline in liver fat on MRI-PDFF is reported.
Time Frame: At week 6
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent change of liver fat
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 8 | 5
Percent change of liver fat | -0.73 (16.272) | 22.07 (27.154)

18. Secondary Outcome: Percentage of Participants Experiencing a Relative Reduction of 30% or Greater of Liver Fat as Assessed by MRI-PDFF
Description: Percentage of participants experiencing a relative reduction of 30% or greater of liver fat as assessed by MRI-PDFF at week 12 are reported.
Time Frame: At week 12
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 8 | 5
Percentage of participants | 25.0 | 0

19. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT)
Description: Change from baseline in ALT is reported.
Time Frame: Baseline, Day 92
Population: The pharmacodynamic (PD) analysis set was to include all participants who received FT-4101 or placebo without major protocol deviations or violations that would have had an impact on PD.
Measure: Least Squares Mean (Standard Error); unit: units per liter (U/L)
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 8 | 5
units per liter (U/L) | -3.0 (6.29) | 40.8 (8.02)

20. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST)
Description: Change from baseline in AST is reported.
Time Frame: Baseline, Day 92
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 8 | 5
U/L | -1.161 (4.2789) | 12.457 (5.4320)

21. Secondary Outcome: Change From Baseline in Gamma-glutamyl Transferase (γGT)
Description: Change from baseline in γGT is reported.
Time Frame: Baseline, Day 92
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 8 | 5
U/L | -2.058 (9.1733) | 46.293 (11.6580)

22. Secondary Outcome: Change From Baseline in Alkaline Phosphatase
Description: Change from baseline in alkaline phosphatase is reported.
Time Frame: Baseline, Day 92
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 8 | 5
U/L | 1.023 (2.2841) | 13.764 (2.8903)

23. Secondary Outcome: Change From Baseline in Total Bilirubin
Description: Change from baseline in total bilirubin is reported.
Time Frame: Baseline, Day 92
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: micromoles per liter (umol/L)
Arm/Group | FT-4101 3.0 mg | Placebo
Number analyzed (Participants) | 8 | 5
micromoles per liter (umol/L) | -0.59 (0.735) | -1.09 (0.932)

24. Secondary Outcome: Maximum Plasma Concentration (Cmax) of FT-4101
Description: Maximum plasma concentration (Cmax) of FT-4101 is reported
Time Frame: Cycle 1 (Day 1), Cycle 4 (Day 14); each Cycle length = 21 days
Population: The pharmacokinetic (PK) analysis set included all participants who received FT-4101 with sufficient evaluable PK concentration data appropriate for the evaluation of interest without major protocol deviations or violations that would have an impact on the absorption, distribution, metabolism, or excretion.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | FT-4101 3.0 mg
Number analyzed (Participants) | 8
nanograms per milliliter (ng/mL)
  Cycle 1 (Day 1) | 62.3 (22.2)
  Cycle 4 (Day 14) | 118 (38.6)

25. Secondary Outcome: Area Under the Concentration-time Curve for a Dosing Interval (AUCtau) of FT-4101
Time Frame: Cycle 1 (Day 1), Cycle 4 (Day 14); each Cycle length = 21 days
Population: Data for this endpoint was not collected and analysed as there were no participants.
Arm/Group | FT-4101 3.0 mg
Number analyzed (Participants) | 0

26. Secondary Outcome: Data for This Endpoint Was Not Collected and Analysed.
Time Frame: Cycle 1 (Day 1), Cycle 4 (Day 14); each Cycle length = 21 days
Population: Data for this endpoint was not collected and analysed as there were no participants.
Arm/Group | FT-4101 3.0 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 20 weeks
Description: The Safety analysis set included all randomized participants who received IP (FT-4101 or placebo) or deuterated water.
Arm/Group | FT-4101 3.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 3/9 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FT-4101 3.0 mg (N=9) | Placebo (N=5)
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was planned for two dosing cohorts (Cohort A and Cohort B), but only Cohort A was included. The study terminated because of observed insufficient efficacy with the studied dose to warrant further investigation. The 3 mg dose didn't raise safety concerns, but to achieve a meaningful result, higher doses would exceed the safe limit based on past studies. Therefore, it was determined that further evaluation of FT-4101 dose escalations for the study indication was not appropriate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT04004325/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT04004325/SAP_001.pdf